CLINICAL TRIAL: NCT06886308
Title: FEASIBILITY and PRELIMINARY EFFICACY of REPETITIVE TRANS-SPINAL MAGNETIC STIMULATION for GAIT RECOVERY AFTER INCOMPLETE SPINAL CORD INJURY
Brief Title: RTsMS and Body Weight-support Treadmill Training After Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Fernanda Natacha Rufino Nogueira, Master in Physical Therapy, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTsMS_BWSTT_iSCI
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: spinal cord injury; gait; body weight- support treadmill training; Repetitive Trans-spinal Magnetic Stimulation; Trans-spinal Magnetic Stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high-frequency rTsMS + BWSTT (Experimental): a randomized, sham-controlled, double-blinded and parallel group trial (10 therapeutic sessions) with the combination between high-frequency rTsMS and body weight-support treadmill training in improving the gait and sensory-motor function of adult patients with chronic incomplete spinal cord injury.
  Interventions: Device: Repetitive trans-spinal magnetic stimulation
- sham rTsMS + BWSTT (Sham Comparator): a randomized, sham-controlled, double-blinded and parallel group trial (10 therapeutic sessions) with the combination between sham rTsMS and body weight-support treadmill training in improving the gait and sensory-motor function of adult patients with chronic incomplete spinal cord injury.
  Interventions: Device: Repetitive trans-spinal magnetic stimulation

INTERVENTIONS:
Device: Repetitive trans-spinal magnetic stimulation — For repetitive trans-spinal magnetic stimulation - rTsMS (high-frequency or sham), volunteers will be positioned comfortably in a lateral decubitus position. High-frequency rTsMS will be applied with an eight-shaped coil over the tenth thoracic vertebra (10 Hz; 100 pulses per train, 20-second interval between trains; 100% resting motor threshold). For sham rTsMS, two coils will be used: (i) a coil connected to the stimulator will be placed behind the patient (away from the spine) to generate the characteristic sound, and (ii) another coil, disconnected from the stimulator, will be placed on the tenth thoracic vertebra. Both real and sham stimulation will last 20 minutes. Gait training with body weight support will be performed on a Biodex Rehabilitation treadmill for 20 minutes. Researchers will assist the patient in foot placement, knee extension, and pelvis/trunk alignment. Body weight support and treadmill speed will be adjusted based on the patient's performance.
  Other Names: Body Weight-support Treadmill Training

SUMMARY:
The aim of this study is to assess the feasibility of combining rTsMS with BWSTT for gait and sensorimotor recovery in individuals with incomplete spinal cord injury.

DETAILED DESCRIPTION:
A randomized, sham-controlled, triple-blinded and parallel group trial (10 therapeutic sessions). Active or sham rTsMS will be combined with body weight-support treadmill training to verify the improvement of gait and sensory-motor function in patients with incomplete spinal cord injury. Assessments will be performed before, after 5 and 10 therapeutic sessions, though: (i) the WISCI-II Index; (ii) ASIA Impairment Scale (AIS), (iii) ASIA Lower Extremities Motor Scale (LEMS), (iv) Ashworth Modified Scale; (v) the Functional Independence Measure (SCIM-III), (vi) the Short Form Health Survey 36 (SF-36) and (vii) the Patient Global Impression of Change Scale - (PGICS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed incomplete spinal cord injury established by a neurologist
* Chronic phase (>1 year)
* 18 and 60 years old, regardless of sex

Exclusion Criteria:

* Community ambulators
* Could not maintain an orthostatic position for 30 seconds without assistance
* Associated neurological and/or orthopedic conditions
* Contraindications for rTsMS
* Diagnosis of cardiac dysfunction, angina, or hemodynamic disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Changes on Walking Index for Spinal Cord Injury II (WISCI-II) | Before the intervention (baseline), after 5 sessions (5 days of intervention) and 10 sessions (10 days of intervention).
  this is international scale, designed to identify an improvement in the ability to perform gait with spinal cord injury under environmental conditions. The WISCI-II is considered standard for gait evaluation of patients with spinal cord injury inserted in clinical trials. The WISCI-II categorizes patients' ability to perform a gait on 20 different levels by considering the following: distance traveled, need for assistance, assistance from others people, and gait devices. The higher the score, the greater the independence in gait.

SECONDARY OUTCOMES:
Changes on ASIA Impairment Scale (AIS) | Before the intervention (baseline), after 5 sessions (5 days of intervention) and 10 sessions (10 days of intervention).
  Sensory-motor function was assessed using the AIS. This assessment measure is part of the guidelines provided by the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI), created by the American Spinal Injury Association. Using the AIS, motor function was measured by the total score of the Upper Extremities Motor Scale (UEMS) and Lower Extremities Motor Scale (LEMS). The UEMS and LEMS are made up of the sum of the strength levels of ten main muscles. Each muscle was given a score ranging from '0' to '5', according to the manual muscle strength assessment scale. Sensory function was measured by the total score of two sensory components assessed in the AIS: 'light touch (LT)' and 'pinprick (PP)'. To assess sensory function, stimuli were applied to the dermatomes as described in the ASIA standardised manuals. The score for each component of the dermatome varies from '0 to 2': 0 = no sensation, 1 = altered sensation and 2 = preserved sensation.
Changes on Spinal cord independence measure (Self-Reported) III - (SCIM-III) | Before the intervention (baseline), after 5 sessions (5 days of intervention) and 10 sessions (10 days of intervention).
  The scale evaluates a patient's ability to perform tasks related to spinal cord injury and tracks improvements in their functional capacity. The SCIM-III scale ranges from 0 to 100 points and is divided into three primary domains: self-care (feeding, bathing, dressing, and hygiene), breathing, sphincter control, and mobility (both indoor and outdoor activities, including transfers). The higher the score on the scale, the greater the functional independence.
Change from Modified Ashworth scale (MAS) | Before the intervention (baseline), after 5 sessions (5 days of intervention) and 10 sessions (10 days of intervention).
  The Modified Ashworth Scale employs a 6-point system to measure the average resistance to passive movement at each joint. In this study, it will assess the following muscle groups: hip flexors and extensors, knee flexors and extensors, and ankle dorsiflexors and plantar flexors. The higher the score on the scale, the greater the degree of spasticity.
Changes on Short-Form Health Survey (SF-36) | Before the intervention (baseline), after 5 sessions (5 days of intervention) and 10 sessions (10 days of intervention).
  The SF-36 is a multidimensional questionnaire consisting of 36 items, encompassed in eight scales or components: i. Functional capacity - 10 items, ii. Limitation by physical resources - 4 items, iii. Pain - 2 items, iv. General health status - 5 items, v. Vitality - 4 items, vi. Social Aspects - 2 items, vii. Limitation by emotional aspects - 3 items, viii. Mental Health - 5 items and one comparative question more for assessment between how current health conditions and a year ago.
Changes on Patient Global Impression of Change Scale - (PGICS) | After 5 sessions (5 days of intervention) and 10 sessions (10 days of intervention).
  The PGICS is a one-dimensional measure in which individuals rate their improvement associated with intervention on a scale of 7 items ranging from "1 = no change" to "7 = Much better". This scale has already been validated in Brazil and has been used in clinical practice assays with spinal cord injury.

CONTACTS AND LOCATIONS:
Overall Officials: Vinicius Cipriano, Student of Physical Therapy, Study Chair — Applied Neuroscience Laboratory
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil